CLINICAL TRIAL: NCT06234514
Title: Traditional Chinese Medicine and Ranibizumab in the Treatment of Macular Cystoid Edema Associated With Retinal Vein Obstruction.
Brief Title: Manage Macular Cystoid Edema With Retinal Vein Obstruction Using Traditional Chinese Medicine and Ranibizumab
Acronym: JQMMT+RA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dongyang People's Hospital (Other)
Responsible Party: Principal Investigator, Zhou Hangshuai, doctor, Dongyang People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JQMMT
Record Dates: First submitted 2024-01-21; First posted 2024-01-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Macular Cystoid Edema
Keywords: Traditional Chinese Medicine; Ranibizumab; Retinal Vein Obstruction
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination Therapy Group (Experimental): During the initial month, the patient consumed Jueling Mingmu decoction daily for one month.
  Patients received monthly intravitreal injections of 0.5mg ranibizumab for the initial three months, followed by additional injections in the subsequent nine months for those who met eligibility criteria.
  Interventions: Drug: Jueling Mingmu decoction; Drug: intravitreal injections of 0.5mg ranibizumab
- Intravitreal Ranibizumab Group (Active Comparator): Patients received monthly intravitreal injections of 0.5mg ranibizumab for the initial three months, followed by additional injections in the subsequent nine months for those who met eligibility criteria.
  Interventions: Drug: intravitreal injections of 0.5mg ranibizumab

INTERVENTIONS:
Drug: Jueling Mingmu decoction — Jueling Mingmu decoction comprises stone cassia, grass cassia, Leonurus, chrysanthemum, red peony, Schizonepeta, poria, plantago, salvia miltiorrhiza, rice bud, licorice. It is designed to clear liver heat, promote diuresis, activate blood circulation, strengthen the stomach, and harmonize spleen functions.
  Arms: Combination Therapy Group
Drug: intravitreal injections of 0.5mg ranibizumab — Patients received monthly intravitreal injections of 0.5mg ranibizumab for the initial three months, followed by additional injections in the subsequent nine months for those who met eligibility criteria.
  Other Names: 0.5mg ranibizumab

SUMMARY:
The objective of this study was to investigate the efficacy and safety of traditional Chinese medicine (Jueling Mingmu Decoction) combined with ranibizumab in the treatment of macular edema with retinal vein obstructive.

DETAILED DESCRIPTION:
Compared to the sole intravitreal injection of ranibizumab, the combined use of traditional Chinese medicine with intravitreal ranibizumab aims to determine if it is more effective in alleviating macular cystoid edema secondary to retinal branch vein occlusion, leading to improved visual prognosis and potentially reducing the frequency of intravitreal drug injections.

ELIGIBILITY:
Inclusion Criteria:

* Foveal center-involved macular edema (ME) lasting less than 9 months
* Central Macular Thickness (CMT) greater than or equal to 250 μm
* Best-Corrected Visual Acuity (BCVA) of 24-73 letters (20/40 to 20/320) in the study eye
* Initial diagnosis with no prior treatments, such as laser therapy or intravitreal injections

Exclusion Criteria:

* Presence of any additional macular pathology, such as age-related macular degeneration (AMD) or diabetic retinopathy (DR) affecting the macula
* Concurrent serious conditions, such as cardiovascular diseases, liver, or kidney diseases
* Concerns or doubts regarding treatment
* Known allergies to the ingredients of the medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Mean number of injections | 48 weeks
  We will calculate the mean number of intravitreal ranibizumab injections at week 48.

SECONDARY OUTCOMES:
Change in BCVA | 48 weeks
  We will assess the participants' best-corrected distance visual acuity by ETDRS charts before and after the treatment at weeks 48.
The mean change of central retinal thickness (CRT). | 48 weeks
  The participants' eyes will be fully dilated; the examiner will take the macular fovea as the center and perform a multi-directional, 6 mm-long, radial linear scan of the most prominent macular lesions and take linear scans in the same direction after the treatment. CRT is defined as the distance between internal limiting membrane and external limiting membrane, excluding the fluid under the retinal pigment epithelium (RPE).

CONTACTS AND LOCATIONS:
Overall Officials: Guangjin Zhao, Study Director — Dongyang People's Hospital
Locations (1):
- Dongyang People's Hospital, Dongyang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No